CLINICAL TRIAL: NCT05164575
Title: Adapting REhabilitation Delivery for Maximum Impact at Home
Acronym: ReDI@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00110340
Record Dates: First submitted 2021-09-16; First posted 2021-12-20 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Osteo Arthritis Knee; Hip Osteoarthritis; Knee Osteoarthritis; Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: eRP-LOw Intensity (eRP-LO) will be an 8-week intervention that includes FOUR virtual visits with a physiotherapist (PT) while eRP-HIgh Intensity (eRP-HI) will be an 8-week intervention with EIGHT virtual weekly visits with a PT. Both interventions will include a progressive resistance exercise program and self-management strategies. Participants will be provided with Theraband to progress exercise intensity, a FitBit to monitor physical activity, an audio-journal to promote self-reflection, and educational materials provided as part of usual OA care.
Who Masked: Outcomes Assessor
Masking Description: ReDI@Home will be a randomized, parallel-arm, single-blind (clinical assessor) feasibility trial with participants randomized to eRP-HI or eRP-LO. An uneven block randomization sequence will be computer-generated with a 1:1 group allocation. Randomization will occur after the pre-intervention visit.
  The research coordinator will randomize participants after the equipment/software set-up and the pre-intervention assessment has been completed. The assigned intervention PT will contact participants to review the eRP and set up appointments as required based on group assignment. We will use one PT for all eRP-LO participants and up to 2 PTs to provide the eRP-HI intervention. Participants will have the same PT throughout, with visits scheduled during the day or early evening at PT and participant preference/availability, as per our previous COACH study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eRP-LOw Intensity (eRP-LO) (Experimental): an 8-week intervention that includes FOUR virtual visits with a physiotherapist
  Interventions: Behavioral: progressive resistance exercise; Behavioral: self-management strategies
- eRP-HIgh Intensity (eRP-HI) (Experimental): an 8-week intervention that includes EIGHT virtual visits with a physiotherapist
  Interventions: Behavioral: progressive resistance exercise; Behavioral: self-management strategies

INTERVENTIONS:
Behavioral: progressive resistance exercise — Progressive resistance exercise program and self-management strategies. Participants will be provided with Theraband to progress exercise intensity, a FitBit to monitor physical activity, an audio-journal to promote self-reflection, and educational materials provided as part of usual OA care.
Behavioral: self-management strategies — Progressive resistance exercise program and self-management strategies. Participants will be provided with Theraband to progress exercise intensity, a FitBit to monitor physical activity, an audio-journal to promote self-reflection, and educational materials provided as part of usual OA care.

SUMMARY:
Hip and knee osteoarthritis (OA) is a burden of disability in adults, with many seeking total joint arthroplasty (TJA) to reduce their symptoms. Almost 50% of people screened for TJA are referred for further rehabilitation rather than TJA. However, access to community-based rehabilitation is limited for those living in rural settings. Recent advances in tele-rehabilitation using smart phone technology, widely available in rural areas, provides a means to access rehabilitation from home.

ReDI@Home will examine the impact of home-based e-Rehabilitation, delivered via smart phone, for rural residents living with moderate to advanced OA. This randomized feasibility trial will compare 2 e-Rehabilitation programs (eRP) of varying intensity (eRP-LOw Intensity [eRP-LO] and eRP-HIgh Intensity [eRP- HI]).

The investigators think that the eRP are feasible and that both eRP will improve OA self-management. However, eRP-HI will improve patient outcomes more than eRP-LO.

DETAILED DESCRIPTION:
ReDI@Home is a randomized feasibility trial that will evaluate implementation of home-based interventions to assist persons with moderate to advanced hip or knee osteoarthritis (OA) living in rural environments with self-management. Although others have used similar web-based interventions for urban patients living with inflammatory arthritis, our selected group of rural residents living with OA, has been under-served with these types of interventions, often due to internet service limitations. Following this feasibility work, a definitive randomized trial of the refined rehabilitation programs relative to usual OA care in rural settings is planned. This feasibility trial is essential before a definitive trial.

Once ReDI@Home is refined and tested, the intervention will be transferable to other provinces/settings where rural residents require rehabilitation. This approach may also work for older adults living in urban areas, whose community rehabilitation access may be limited due to physical distancing associated with COVID-19.

Objectives and Hypotheses

ReDI@Home will examine the impact of home-based e-Rehabilitation, delivered using smart phone technology, for those living with moderate to advanced OA who reside in rural regions. This randomized feasibility trial will compare 2 e-Rehabilitation Programs (eRP):

eRP-LOw Intensity (eRP-LO) will be an 8-week intervention that includes FOUR virtual visits with a physiotherapist (PT) while eRP-HIgh Intensity (eRP-HI) will be an 8-week intervention with EIGHT virtual weekly visits with a PT. Both interventions will include a progressive resistance exercise program and self-management strategies. Participants will be provided with Theraband to progress exercise intensity, a FitBit to monitor physical activity, an audio-journal to promote self-reflection, and educational materials provided as part of usual OA care.

ReDI@Home will answer the following research questions:

1. Are eRP using smart phone technology feasible for rural Albertans living with moderate to advanced OA?
2. If feasible

   1. are eRP effective?
   2. do eRP vary in effectiveness based on intensity and participant characteristics?

1. Feasibility will evaluate:

1. Participant recruitment/participation/retention/satisfaction
2. Treatment fidelity (delivery of eRP as intended): will be compared within and between groups.
3. Outcomes/Outcome measure utility and responsiveness 2. Effectiveness will compare

a. Patient outcomes between the 2 interventions using validated measures: i. Self-management (primary effectiveness outcome) using the Patient Activation Measure ii. Lower extremity strength/balance using the 30-second Chair Stand test iii. Pain and Function using the Hip disability and Osteoarthritis Outcome Score(HOOS)/Knee Osteoarthritis Outcome Score(KOOS) and Intermittent and Constant Osteoarthritis Pain (iCOAP) score iv. Physical activity and the Sedentary Lifestyle Index(SLI) using FitBit-measured step count v. Change from pre-intervention using Global Rating of Change vi. Anxiety/depression using the Hospital Anxiety and Depression Scale (HADS) vii. Pain catastrophizing using the Pain Catastrophizing Scale (PCS) viii. Social Support, Network, & Participation using the Canadian Longitudinal Study of Aging (CLSA) ix. Health literacy using the Health Literacy Questionnaire (HLQ) b. Responders versus non-responders in both eRP to refine selection criteria/eRP content The investigators hypothesize that the eRP will be feasible and that both eRP will improve OA self-management, but there may be non-responders in both eRP. eRP-HI will improve all patient outcomes more than eRP-LO.

Research Method/Procedures DESIGN: ReDI@Home will be a randomized, parallel-arm, single-blind (clinical assessor) feasibility trial with participants randomized to eRP-HI or eRP-LO. An uneven block randomization sequence will be computer-generated with a 1:1 group allocation. Randomization will occur after the pre-intervention visit.

SCREENING: For feasibility, the investigators will determine the number of patients eligible for participation as well as the reason for ineligibility (e.g., metro Edmonton residence, technology issues &/or data limitations, etc.). For those eligible, but who refuse participation, reasons for refusal including apprehension with technology or privacy (e.g., having virtual video home visits with PT) will be noted. The investigators will also complete semi-structured interviews with this sub-group (See Qualitative Assessment below). Feasibility outcomes will determine the a) reach of eRP in rural areas and b) rural residents' willingness to participate in such programs. The semi-structured interviews with those refusing to participate are anticipated to be shorter in duration, 20-30 minutes. These interviews will be with those who are willing via the phone or Zoom. All interviews will be scheduled at a time convenient for the interviewer and the participant. The meetings will be set up over email or the phone and take place on Zoom or on the phone, whichever is better for the participant.

ENROLLMENT: Enrollment will occur during the Camrose- or Edmonton-based surgical eligibility clinic visit. Clinic staff will identify eligible patients (using the referral to identify diagnosis of OA and patient address for rural residence) and determine if they wish to talk to researchers. If the research personnel is in attendance at these clinics they will confirm eligibility, explain the study and obtain signed consent (electronic format: e-consent) from eligible volunteers. When the research personnel is not in attendance, clinic staff will determine the patients' interest in talking to researchers and will obtain their contact information using the 'consent to contact form' to pass on to the researchers. Researchers will contact patients by telephone and obtain e-consent from eligible and willing participants. For potentially eligible participants completing virtual appointments due to COVID-19, clinic staff will determine their interest in talking to researchers and will obtain the patients' contact information via phone using the 'consent to contact script' to pass on to the researchers. Researchers will contact patients by telephone and obtain e-consent from eligible and willing participants.

All participants will receive written information regarding OA management/exercises provided by the intake clinics as per usual care. They will receive a tripod to hold their smart phone/tablet, a Fitbit, and 2 Therabands of varying intensity. Research personnel will register and install the Fitbit, YARO avatar, and Zoom for Health 'apps' on participants' smart phones/tablets along with video instructions on their use; there are no costs for these apps.

For those enrolled virtually, these same items will be mailed with instruction sheets. The research coordinator will phone the participants once items are received and help them to install the apps and setup their Fitbit, YARO avatar and Zoom for Health. The investigators previously completed Fitbit setup successfully using mailed instructions (with a YouTube link) in a similar patient group (post-TJA) with phone assistance as needed.

Although all participants will be encouraged to use the planned smartphone technology (and only be enrolled if they meet the technology eligibility criteria), as a feasibility trial, the investigators must plan for failure of the intervention technology delivered as intended in some cases. If such failure occurs (including unwillingness of patients to continue with the intervention technology), the investigators will adapt intervention delivery and research assessment to be web- or telephone-based to retain participants in the eRPs and research evaluation. Change in eRP delivery mode is included in the feasibility assessment.

RESEARCH ASSESSMENT: A research associate who is not engaged with the intervention and blinded to group allocation will contact participants using secured Zoom for Health at 0-weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization to complete the standardized measures. At the pre-intervention assessment, socio-demographics, co-morbidities, and employment status will be collected. The 30-second Chair Stand test will only be completed if it can be done safely. Participants will connect via Zoom for Health after receiving an embedded link in an email sent by the assessor. All data will be stored on the remote secure server, not the assessor's tablet.

Participants will wear the Fitbit for 10 weeks (i.e., one- week before and during the intervention period) and then again for at least 1 week before the 6- and 12-month assessments, to measure step count- derived physical activity and SLI using their Fitbit Dashboard.

RANDOMIZATION: The research coordinator will randomize participants after the equipment/software set-up and the pre-intervention assessment has been completed. The assigned intervention PT will contact participants to review the eRP and set up appointments as required based on group assignment. The investigators will use one PT for all eRP-LO participants and up to 2 PTs to provide the eRP-HI intervention. Participants will have the same PT throughout, with visits scheduled during the day or early evening at PT and participant preference/availability, as per our previous COACH study.

INTERVENTION: Both eRPs will be led by PTs experienced in working with patients with hip/knee OA. Participants will attach their cellphone/tablet to the tripod selfie-stick provided at enrollment. They will receive an embedded link in an email that will connect them to a secure Zoom for Health session. The link will also connect their camera, cell phone/tablet microphone and speaker to the eRP providers' tablet. Sessions will be recorded with data stored on a secure server along with the Kinetisense data to allow assessment of change in function and gait over time as well as treatment fidelity. Both eRP will have the following components: Progressive Exercises will include an evidence-based progressive resistance training program using Theraband and bodyweight, with weekly (eRP-HI) or biweekly (eRP-LO) progression. PTs will use Kinetisense to observe exercises/gait performance and progress exercise intensity as tolerated, encouraging exercise completion at least 1-2 times between PT sessions. Self-management will include a) physical / mental / emotional self-management, and b) exercise / physical activity advice to enhance uptake. Physical activity, using the Fitbit will be measured by daily step count and energy expenditure; our recent work found that Fitbit step count and energy expenditure correlate well with a research grade accelerometer. Daily audio-journaling using YARO as an adjunct to PT interactions will promote self-reflection for mental health, encourage healthy lifestyle choices (e.g., diet, sleep, physical activity) as well as exercise compliance using a daily query about exercise performance (informal exercise log through self-report). The screening clinics' educational materials, including exercise booklets, will be provided as part of usual care.

eRP-Lo will include 4 sessions over 8 weeks while eRP-HI will include 8 sessions over 8 weeks, with each session lasting ~45-60 minutes. At each visit, the PT will discuss OA self-management and review and progress exercise performance. PTs will individualize exercises to patient tolerance (i.e., patients will exercise at different intensities and progress as able) and the home environment. Delivery of the self-management content will be prioritized by the participant and PT, so that discussions focus on each participant's individual needs to personalize the approach. PTs will also encourage a) physical activity using the Fitbit as an aid to set activity goals and b) audio-journaling with YARO for self-reflection. Participants will be encouraged to exercise, increase physical activity, audio-journal and/or access educational materials between sessions using individual goal-setting to promote patient activation.

Up to 20 eligible participants WHO REFUSE PARTICIPATION will be given an option to participate in a brief semi-structured interview to understand their attitudes, perceptions, and interest in participating in eRP; understanding the barriers to participation may allow refinement of the eRP improve their reach. A 'Quality of Experience' assessment will be completed with up to 20 eligible participants WHO COMPLETE THE eRPS AND PT PROVIDERS (N= 3-5) using semi-structured interviews to understand perceptions of program value, appropriateness, effectiveness, acceptability and satisfaction with the eRPs. Twenty participants from each of these populations should allow us to reach data saturation. An experienced qualitative assessor working on Tele-Rehab 2.0 will complete all interviews; this assessor is independent of eRP delivery. Interviews will be recorded and field notes (impressions noted by the interviewer), will be analyzed thematically and inductively to identify ideas, categories and themes of interest. Qualitative data will further inform eRP refinement.

In addition to the validated outcome measures, the investigators will also collect the following information at the pre- intervention interview to evaluate how patient characteristics impact eRP outcomes:

* Demographics (e.g. age, sex)
* Affected joint (hip or knee)
* Comorbidities using the validated Canadian National Population Health Survey listing, including obesity (BMI), and socio-demographics.
* Occupation (e.g. employed, retired, other)
* Living Arrangements (e.g. lives alone or with others; relationship with participant)
* Residence location (e.g. small town, farm) SAMPLE SIZE: Considering 2 groups evaluated over 4 time-points, small to medium effect size (d=0.3), moderate correlation (r=0.4) and allowing 15% attrition, the investigators will enroll 120 participants (n=60/group).

ELIGIBILITY:
Inclusion Criteria:

* Present to the Edmonton or Camrose screening clinic with moderate to advanced hip or knee OA not eligible for TJA within one year (i.e., not RA, not currently waiting for TJA)
* Reside outside of metro Edmonton (defined by StatsCan)
* Access to a smart phone or tablet with embedded camera that can accept intervention software, with a current data plan in place and/or strong WiFi or ethernet connection*
* English-speaking
* Are in need of guided exercise but are a functional community ambulator (with or without aids)
* Experience hip or knee pain multiple days a week
* Have activity limitations because of joint pain

Exclusion Criteria:

* Patients who are not eligible for TJA due to uncontrolled medical conditions (e.g., diabetes, hypertension) will be excluded due to safety concerns (i.e., undertaking exercise in their health state).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Change in Patient Activation Measure from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  Self-management A13-item survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare.
  PAM segments individuals into one of four activation levels along an empirically derived 100-point scale. Each level provides insight into an extensive array of health-related characteristics, including attitudes, motivators, and behaviors. Individuals with a low score do not yet understand the importance of their role in managing their own health, and have significant knowledge gaps and limited self-management skills. Individuals with higher scores are proactive with their health, have developed strong self management skills, and are resilient in times of stress or change.

SECONDARY OUTCOMES:
Change in Hip Disability and Osteoarthritis Outcome Score from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  Measures pain, other symptoms, activities of daily living, sports/recreation, and hip-related quality of life The outcome score consists of 40 items assessing 5 subscales. The 5 separate patient-relevant dimensions are Pain (P), Symptoms (S), Activity limitations daily living (ADL), Function in sport and recreation (SP) and hip related quality of life (QOL) P includes 10 items with a total score of 40 points, S includes 5 items with a total score of 20, ADL includes 17 items with a total score of 68, and SP and QOL include 4 items with a total score of 16 each.
  For each question, standardized answer options are given in 5 Likert-boxes with scores from 0 to 4 (no, mild, moderate, severe and extreme). To interpret the score, the outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms
Change in Knee Osteoarthritis Outcome Score from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  A validated, self- administered questionnaire measuring knee pain, stiffness, daily activity, sports/recreation, and quality of life in people with knee OA, with known clinically meaningful change.
  The five patient-relevant subscales of KOOS are scored separately: Pain (nine items), Symptoms (seven items), ADL Function (17 items), Sport and Recreation Function (five items), and Quality of Life (four items) A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems. An aggregate score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately.
Change in Intermittent and Constant Osteoarthritis Pain from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  A measure that evaluates pain related to hip or knee OA. 11-item tool is designed to assess pain in individuals with hip or knee osteoarthritis taking into account both constant and intermittent pain experiences. There are two versions of this tool; one to assess pain in the knee joint and another assessing pain in the hip joint.
  There are 11 items on the questionnaire. Items are numbered according to the order they appear in the questionnaire.
  Items are scored from 0 to 4 as follows:
  Items 1, 2, 3, 4, 5, 6, 8, 9, 10, 11 0 = not at all/I don't have <constant pain/pain that comes and goes>
  1. = mildly
  2. = moderately
  3. = severely
  4. = extremely Item 7
  0 = never/I don't have <constant pain/pain that comes and goes>
  1. = rarely
  2. = sometimes
  3. = often
  4. = very often
  High scores (scores closer to 44) indicate worse pain.
Change in Hospital Anxiety and Depression Scale from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  a valid and reliable questionnaire that includes 14 items (7 depression-related items and 7 anxiety-related items) will evaluate if depressive and/or anxiety symptomology, common in this group, is present, determine the impact of eRP on symptomology if present.
  Scores of less than 7 indicate non-cases 8-10 Mild 11-14 Moderate 15-21 Severe
Change in Pain Catastrophizing Scale from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  Assesses distress, negative cognitive & emotional responses to actual or anticipated pain.
  13 statements describing different thoughts and feelings that may be associated with pain. Users indicate the degree to which they have these thoughts and feelings when they are experiencing pain, with 0 being not at all and 4 being all the time. A maximum score of 52 and a minimum score of 0, with higher scores indicating pain catastrophizing. A total PCS score of 30 represents clinically relevant level of catastrophizing. A total PCS score of 30 corresponds to the 75th percentile of the distribution of PCS scores in clinic samples of chronic pain patients
Change in Global Rating of Change from baseline to post intervention and 6-months and 12-months | At 9-weeks (post-intervention) and 6- and 12-months following randomization.
  Completed post-intervention by all participants and e-Rehabilitation Program (eRP) providers assessing self-reported (participant) or provider (eRP PT) change from pre-intervention.
  4 questions. Scoring options of "Much better [+3], Better [+2], Somewhat better [+1], Same [0], Somewhat worse [-1], Worse [-2], Much worse [-3]" AND "Very satisfied [+3], Satisfied [+2], Somewhat satisfied [+1], Neutral [0], Somewhat dissatisfied [-1], Dissatisfied [-2], Very dissatisfied [-3]" Range from -12 to +12. Minimum value: -12 Maximum value: +12 Higher scores indicate greater positive change and higher satisfaction. Lower scores indicate lower positive change and lower satisfaction.
Change in 30-second Chair Stand test from baseline to post intervention and 6-months and 12-months | At 0- weeks (pre-intervention), 9-weeks (post-intervention) and 6- and 12-months following randomization.
  Measure of lower extremity strength/balance. records the number of times a participant can stand and sit in a chair in 30 seconds. It is a valid tool to assess people with hip or knee OA, with a minimally clinical difference of 1.64
Change in Sedentary Lifestyle Index and Physical Activity from baseline to post intervention and 6-months and 12-months | At 9-weeks (post-intervention) and 6- and 12-months following randomization.
  Using FitBit step count we will determine the SLI (<5000 or >/=5000 steps/day) to evaluate the e-Rehabilitation Program's impact on stationary behavior. Increase in physical activity by 2,000-2,500 steps per day is reported to improve health outcomes, but even small changes in activity levels have been associated with health benefits
Canadian Longitudinal Study of Aging | At screening/enrollment
  A social support questionnaire that asks about the support that is available to the individual. Social Network questionnaire asks about the people who live in one's household and their relationship. Social participation questionnaire asks about the individual's social activities.
  CLSA includes measures that cover both structural (e.g., social network size, frequency of contact) and functional (perception of support received) domains relevant to social support. The CLSA Questionnaire includes 15 items pertaining to the respondent's social network; these items include marital/partner status, living arrangements, family composition, social ties and social contacts.
  Higher scores indicate greater levels of social support. The investigators will describe this in the feasibility trial.
Health Literacy Questionnaire | At screening/enrollment
  To assess the needs and challenges of a wide range of people in the community. Number of items: 44 Items are scored from 1-4 in the first 5 scales (Strongly Disagree, Disagree, Agree, Strongly Agree), and from 1-5 in scales 6-9 (Cannot Do, Very Difficult, Quite Difficult, Easy, Very Easy).
  Minimum 44 Maximum 197

CONTACTS AND LOCATIONS:
Locations (1):
- Edmonton Bone and Joint Centre, Edmonton, Alberta, Canada